CLINICAL TRIAL: NCT01790997
Title: The Role of DLBS1033 in Evaluating Bleeding Profile and Clinical Outcome in Patients With Acute Ischemic Stroke: Comparison With Aspirin and Clopidogrel
Brief Title: Efficacy of DLBS1033 in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-UST-001.11
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-01

CONDITIONS: Acute Ischemic Stroke
Keywords: DLBS1033; Lumbrokinase; Acute ischemic stroke; Bleeding profile; Clinical outcome; Aspirin; Clopidogrel
MeSH Terms: conditions — Ischemic Stroke | interventions — DLBS 1033; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment I (Experimental): 1 tablet of DLBS1033 490 mg thrice daily, after meal
  Interventions: Drug: DLBS1033
- Treatment II (Active Comparator): 1 tablet of aspirin 80 mg once daily, after meal
  Interventions: Drug: Aspirin
- Treatment III (Active Comparator): 1 tablet of clopidogrel 75 mg once daily, after meal
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: DLBS1033 — 1 tablet of DLBS1033 490 mg thrice daily, after meal
  Arms: Treatment I
Drug: Aspirin — 1 tablet of aspirin 80 mg once daily, after meal
  Arms: Treatment II
Drug: Clopidogrel — 1 tablet of clopidogrel 75 mg once daily, after meal
  Arms: Treatment III

SUMMARY:
This is a 3-arm, prospective, randomized, double-blind, and controlled clinical study, with 3 months of treatment to evaluate efficacy of DLBS1033 in bleeding profile and clinical outcome in patients with acute ischemic stroke compared with aspirin and clopidogrel, as active controls.

DETAILED DESCRIPTION:
There will be 3 groups of treatment; each group will consist of 43 subjects with the treatment regimens :

* Treatment I : 1 tablet of DLBS1033 490 mg thrice daily, after meal
* Treatment II : 1 tablet of aspirin 80 mg once daily, after meal
* Treatment III : 1 tablet of clopidogrel 75 mg once daily, after meal

Bleeding profile (by measuring INR value, PT, and aPTT) and clinical outcome (by measuring Gadjah Mada Stroke Scale and Barthel Index) to evaluate the efficacy of the investigational drug will be performed at baseline and end of study (Month 3rd). General condition of the subjects will be followed-up every month over three months of study medication.

Physiotherapy will be provided to the subjects by the assigned Physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 20-80 years old
* Having non-bleeding stroke in CT scan examination
* Having stroke attack onset ≤ 96 hours
* Living in 100 km from RSUP Dr Sardjito Jogjakarta

Exclusion Criteria:

* Having recurrence stroke
* Having Transient Ischemic Attack (TIA)
* Have been regularly taking anti-aggregation agent
* Having intracerebral and subarachnoid bleeding stroke
* Subjects and their family do not know when the stroke symptoms appeared
* History of haemostasis disorder
* History of or will have surgery within 6 months prior to screening

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in INR value | 3 Months
  Change in INR (international normalized ratio) value from baseline to end of study (Month 3rd)

SECONDARY OUTCOMES:
Change in PT | 3 Months
  Change in PT (prothrombin time) from baseline to end of study (Month 3rd)
Change in aPTT | 3 Months
  Change in aPTT (activated-partial thromboplastin time) from baseline to end of study (Month 3rd)
Change in Gadjah Mada Stroke Scale | 3 Months
  Change in Gadjah Mada Stroke Scale from baseline to end of study (Month 3rd)
Change in Barthel Index | 3 Months
  Change in Barthel Index from baseline to end of study (Month 3rd)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Setyopranoto, dr., SpS(K), Principal Investigator — Stroke Unit, Department of Neurology, Faculty of Medicine, Gadjah Mada University, dr. Sardjito Hospital, Jogjakarta, Indonesia
Locations (1):
- Stroke Unit, Department of Neurology, Faculty of Medicine, Gadjah Mada University, dr. Sardjito Hospital, Yogyakarta, Jogjakarta, Indonesia